CLINICAL TRIAL: NCT05251805
Title: Phase I Clinical Trial Evaluating the Safety and Feasibility of Bone Marrow Aspiration From Ribs During Thoracic Surgery
Brief Title: The Safety and Feasibility of Costal Bone Marrow Aspiration During Thoracic Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Initial observations suggest challenges in performing bone marrow aspiration in the first few patients enrolled in the study.
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UZB-DVH-2022-01
Record Dates: First submitted 2022-01-27; First posted 2022-02-23 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-04

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Costal bone marrow aspiration (Experimental): 4 NSCLC patients undergoing surgery from which blood samples, bone marrow aspirate and lung tumor tissue will be collected
  Interventions: Procedure: Blood, bone marrow and lung tumor tissue collection

INTERVENTIONS:
Procedure: Blood, bone marrow and lung tumor tissue collection — Blood sampling: 12ml of blood will be collected during the routine pre-operative blood collection
  Bone marrow aspiration during thoracic surgery: following the surgical intervention, bone marrow aspiration will be performed through the incisions made for the thoracic procedure. The ribs lying directly above and below the trocar incision will be exposed. A bone marrow needle will be advanced into the periost until the needle tip reaches the bone marrow. After removing the stylet a 2ml syringe will be attached to the aspiration needle and 0.5ml to 2ml of bone marrow will be aspirated before removing the needle. This procedure will be repeated twice for every trocar site, for a maximum of 3 trocar sites, or until 5ml of bone marrow aspirate is obtained.
  Lung tumor collection: all surgical samples will be analyzed by our anatomopathological department. Viable and fresh material, not used for the diagnostic purposes, will be sent to the LMCT.

SUMMARY:
This pilot trial is designed to evaluate the feasibility and safety of obtaining bone marrow from costal aspiration during surgery.

The investigators hypothese that sufficient bone marrow-derived HSPC's (which represent only 0,1% of the total bone marrow fraction) can be derived by rib bone marrow aspiration for ex vivo single-cell evaluation, optimization of a 3D BMN platform and preclinical ex/in vivo assessment in patient-derived organoids and murine xenograft models.

DETAILED DESCRIPTION:
This pilot trial is designed to evaluate the feasibility and safety of obtaining bone marrow from costal aspiration during surgery.

Previous trials demonstrated the feasibility of micro-metastasis detection in rib marrow aspirate. This procedure appears safe since no adverse events were documented during previous trials. The investigators hypothesize this technique can be used to obtain sufficient bone marrow-derived HSPC's (which represent only 0,1% of the total bone marrow fraction) for ex vivo single-cell evaluation, optimization of a 3D BMN platform and preclinical ex/in vivo assessment in patient-derived organoids and murine xenograft models. The use of rib marrow eliminates the need for extra incisions because the cuts made for trocar placement or the thoracotomy can be re-used. Therefore, the investigators hypothesize that the patients undergoing costal bone marrow aspiration during surgery will not experience extra discomfort. Every patient undergoing thoracic surgery is treated according to ERAS protocols with a major emphasis on pain control.

If the feasibility and safety of bone marrow aspiration are confirmed by this pilot trial, the investigators plan to conduct a large-scale study in which they will collect and bank blood, bone marrow and tumor per NSCLC patient. With this unique autologous biological material collection, the investigators aspire to conduct innovative research into the current resistance mechanisms of NSCLC to immunotherapy;

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing thoracic surgery for a confirmed or suspected lung cancer

Exclusion Criteria:

* Uncertainty of pre-operative diagnosis, exception is per-op frozen section analysis confirming malignity
* ASA ≥ 3
* Bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Costal Bone Marrow Aspiration: 10 NSCLC patients undergoing surgery from which blood samples, bone marrow aspirate and lung tumor tissue will be collected
  Blood, bone marrow and lung tumor tissue collection: Blood sampling: 12ml of blood will be collected during the routine pre-operative blood collection
  Bone marrow aspiration during thoracic surgery: following the surgical intervention, bone marrow aspiration will be performed through the incisions made for the thoracic procedure. The ribs lying directly above and below the trocar incision will be exposed. A bone marrow needle will be advanced into the periost until the needle tip reaches the bone marrow. After removing the stylet a 2ml syringe will be attached to the aspiration needle and 0.5ml to 2ml of bone marrow will be aspirated before removing the needle. This procedure will be repeated twice for every trocar site, for a maximum of 3 trocar sites, or until 5ml of bone marrow aspirate is obtained.
  Lung tumor collection: all surgical samples will be analyzed by our anatomopathological department. Viable and fresh material, not used for the diagnostic purposes, will be sent to the LMCT.
Period: Overall Study
Arm/Group | Costal Bone Marrow Aspiration
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Costal Bone Marrow Aspiration
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 4

OUTCOME MEASURES:

1. Primary Outcome: The Occurrence of Adverse Events Following Costal Bone Marrow Aspiration Classified by Calvien Dindo
Description: All adverse events will be classified by the Clavien Dindo classification. The study will be closed prematurely if 2 patients experience a grade 3 adverse event directly related to the bone marrow aspiration
Time Frame: 7 days following surgery
Measure: Mean (Full Range); unit: total of adverse events
Arm/Group | Costal Bone Marrow Aspiration
Number analyzed (Participants) | 4
total of adverse events | 6 [2 to 11]

2. Secondary Outcome: Measurement of the Amount of HPSC's That Can be Obtained From Costal Bone Marrow
Description: a minimum of 2x106 Lin- CD34+ HPSC are required to allow single cell sequencing, 3D bone marrow cultivation and transplantation in immunodeficient mice.
Time Frame: 7 days following aspiration from the bone marrow
Population: the HPSC's couldn't be measured as the bone marrow aspiration stayed unsuccesfull. hPSC's needed to be extracted from the costal bone marrow. However, since the bone marrow aspiration from the costal bone marrow stayed unsuccesfull, no hPSC's could be extracted and thus the amount could not be measured.
Groups:
- Costal Bone Marrow Aspiration: 4 NSCLC patients undergoing surgery from which blood samples, bone marrow aspirate and lung tumor tissue will be collected
  Blood, bone marrow and lung tumor tissue collection: Blood sampling: 12ml of blood will be collected during the routine pre-operative blood collection
  Bone marrow aspiration during thoracic surgery: following the surgical intervention, bone marrow aspiration will be performed through the incisions made for the thoracic procedure. The ribs lying directly above and below the trocar incision will be exposed. A bone marrow needle will be advanced into the periost until the needle tip reaches the bone marrow. After removing the stylet a 2ml syringe will be attached to the aspiration needle and 0.5ml to 2ml of bone marrow will be aspirated before removing the needle. This procedure will be repeated twice for every trocar site, for a maximum of 3 trocar sites, or until 5ml of bone marrow aspirate is obtained.
  Lung tumor collection: all surgical samples will be analyzed by our anatomopathological department. Viable and fresh material, not used for the diagnostic purposes, will be sent to the LMCT.
Arm/Group | Costal Bone Marrow Aspiration
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: all adverse events were captured from signing the ICF till 30 days post surgery
Arm/Group | Costal Bone Marrow Aspiration
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Costal Bone Marrow Aspiration (N=4)
Nausea (Gastrointestinal disorders) | 3 (4)
injection site reaction (Infections and infestations) | 1 (1)
Hypoxia (Blood and lymphatic system disorders) | 2 (5)
hypokalemia (Blood and lymphatic system disorders) | 1 (1)
fever (General disorders) | 1 (1)
hypotension (Blood and lymphatic system disorders) | 2 (2)
constipation (Gastrointestinal disorders) | 1 (1)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
phlebitis (Blood and lymphatic system disorders) | 1 (1)
itchy back (General disorders) | 1 (1)
sleeplessness (General disorders) | 1 (1)
stomach ache (Gastrointestinal disorders) | 1 (1)
stress (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT05251805/Prot_000.pdf